CLINICAL TRIAL: NCT02074163
Title: ASIS for Botox in Chronic Migraine
Acronym: ASISinCM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASIS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCTNS088800; R01NS088800 (Other Grant/Funding Number: NATIONAL INSTITUTE OF NEUROLOGICAL DISORDERS AND STROKE)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Migraine More than15 Days Per Month, and Lasting 4 Hours a Day or Longer.
Keywords: Subdermal bloodless space; Subdermal injection; injectable EMG needle; electrical stimulation; MRI with Gadolinium; Chronic Migraine; intramuscular injection
MeSH Terms: interventions — Gadolinium; Gadolinium DTPA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (19):
- Glabella (Experimental): Glabella
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Frontal (Experimental): Frontal
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Temporal (Experimental): Temporal
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Occipital (Experimental): Occipital
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Paraspinal (Experimental): Paraspinal
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Trapezius (Experimental): Trapezius
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Change in frequency of headache days (Experimental): Change in frequency of headache days as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30.
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24,; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change in hrs of HA on HA days (Experimental): Change in hrs of HA on HA days as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30.
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24,; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Adverse Reactions with Facial paresis (Experimental): Facial paresis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Eyelid ptosis (Experimental): Eyelid ptosis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Bronchitis (Experimental): Bronchitis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Neck pain (Experimental): Neck pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle stiffness (Experimental): Musculoskeletal stiffness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscular weakness (Experimental): Muscular weakness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Myalgia (Experimental): Myalgia as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle pain (Experimental): Musculoskeletal pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle spasms (Experimental): Muscle spasms as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions Injection site pain (Experimental): Injection site pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Hypertension (Experimental): Hypertension as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally

INTERVENTIONS:
Drug: Gadolinium — Gadolinium .1cc/ diluted with .9ccNS intramuscularly with ASIS Device for 30 patients. Total cumulative Persistent % of Gadolinium intramuscularly on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Frontal; Glabella; Occipital; Paraspinal; Temporal; Trapezius
Drug: Gadolinium — Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium intramuscularly on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Frontal; Glabella; Occipital; Paraspinal; Temporal; Trapezius
Drug: Efficacy of Botox intramuscularly at Week 6 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 6, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox intramuscularly at Week 12 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 12, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox intramuscularly at Week 18 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 18, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox intramuscularly at Week 24, — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 24, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox intramuscularly at Week 30 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 30, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox subdermally at Week 6 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 6, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox subdermally at Week 12 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 12, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox subdermally at Week 18 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 18, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox subdermally at Week 24 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 24, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Efficacy of Botox subdermally at Week 30 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 30, in terms of Change in frequency of headache days, and Change in hrs of HA on HA days.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change in frequency of headache days; Change in hrs of HA on HA days
Drug: Adverse Reactions of Botox intramuscularly — Adverse Reactions of Botox (onabotulinumtoxinA) intramuscularly at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain
Drug: Adverse Reactions of Botox subdermally — Adverse Reactions of Botox (onabotulinumtoxinA) subdermally at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain

SUMMARY:
Botox acts on nerve endings, yet there are no nerve endings inside the muscle, where they are typically injected. All nerves terminate on the fascia, where ASIS device can precisely deliver Botox by creating that subdermal bloodless space, between the skin and muscle. Thus enhancing and prolonging Botox's efficacy, at the same time prevent it's unnecessary adverse reactions and distant spread, especially since Botox has no reason to travel to the rest of the body any way.

DETAILED DESCRIPTION:
Aim 1 over 6 months will demonstrate ASIS device's consistent performance on 60 adult subjects with Chronic Migraine (≥15 days per month, with headache lasting 4 hours a day or longer). Gadolinium will be injected with ASIS subdermally (30) or conventional intramuscularly (30) for these 6 muscle groups: Glabella, Frontal, Temporal, Occipital, Paraspinal, and Trapezius. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. Since there isn't a way to measure level of Gadolinium within it, or any other (e.g. Botox) for that matter, at least the Prolongation of Gadolinium may be approximated by the greater or longer Persistent % on MRI. However, this approximation can only work if the variables are minimized to the same population with Chronic Migraine, and these particular 6 muscle groups. Case in point, patients with Chronic Migraine presumably have hyperactive Glabella, Frontal, Temporal, Occipital, Paraspinal, and Trapezius muscles, so expectantly will have shortened Gadolinium intramuscularly Persistent %, and somewhat Gadolinium subdermally Persistent % as well due to agitation, thus these Persistent % values in Chronic Migraine patients will not be like those of normal patients, or even the same between these 6 different muscle groups. Therefore, the Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, will be specific and valuable indicators to help us modify the Botox dosage and duration to inject into that "unknown" subdermal bloodless space for Aim 2.

Aim 2 over 12 months, using Botox, instead of Gadolinium, to demonstrate the advantages of ASIS device subdermally over intramuscularly, for the particular 6 muscle groups on the same 60 Chronic Migraine adults. Given that there isn't a way to detect Botox in the peripheral blood to document Prolongation of Botox Pharmacokinetically, this Relative Prolongation Ability is our best and only possible way to demonstrate that subdermal bloodless space's ability on Botox. Although valuable, that Relative Prolongation Ability Score from Aim 1 isn't absolutely required to start Aim 2. Hypothetically speaking, if that subdermal bloodless space in patients with e.g., Chronic Migraine somehow failed to show prolongation of half-life for Gadolinium in Aim 1, we can still proceed with primary interest being therapeutic comparison for Botox in Aim 2, in terms of reduction in Number of Headache Days from Baseline, and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Must have history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society for at least 3 months prior to enrollment.
* Must be able to understand the requirements of the study including maintaining a headache diary, and signing informed consent.
* If taking migraine preventive, must be on a stable dose of preventive medication for at least 3 months.

Exclusion Criteria:

* Has headache disorders outside IHS-defined chronic migraine definition.
* Has evidence of underlying pathology contributing to their headaches.
* Has any pathology of the salivary glands such as sialadenitis (e.g. Sjogren's syndrome, viral or bacterial sialadenitis) or condition or symptom that would alter the content of saliva.
* Has any medical condition that may increase their risk with exposure to Botox including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.
* Has profound atrophy or weakness of muscles in the target areas of injection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative Prolongation Ability Score for Gadolinium subdermally injected. | 12 months
  Gadolinium will be injected with ASIS subdermally (30) or conventional intramuscularly (30) in Chronic Migraine adult patients for these 6 muscle groups: Glabella, Frontal, Temporal, Occipital, Paraspinal, and Trapezius. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. This approximation can only work if the variables are minimized to the same population with Chronic Migraine, and these particular 6 muscle groups. The Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, in Chronic Migraine patients will not be like those of normal patients, or even the same between these 6 different muscle groups, but valuable indicators to help us modify Botox dosage and duration to inject into "unknown" subdermal bloodless space for Aim 2.

SECONDARY OUTCOMES:
Efficacy of Botox intramuscularly vs. subdermally in Chronic Migraine. | 12 months
  Efficacy of Botox intramuscularly vs. subdermally with ASIS Device at Week 6,12,18, 24, and 30; in terms of Change from baseline in frequency of headache days, and Change from baseline in total cumulative hours of headache on headache days.

OTHER OUTCOMES:
Adverse Reactions of Botox intramuscularly vs. subdermally in Chronic Migraine. | 12 months
  Adverse Reactions of Botox intramuscularly vs. subdermally:
  Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Li Nguyen, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM INC; Thanh Phung, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM, INC
Locations (1):
- Automatic Subdermal Injector System, Inc, Westminster, California, United States

REFERENCES:
- [Background] Bartleson JD, Cutrer FM. Migraine update. Diagnosis and treatment. Minn Med. 2010 May;93(5):36-41. PMID 20572569
- [Background] Lorenc ZP, Kenkel JM, Fagien S, Hirmand H, Nestor MS, Sclafani AP, Sykes JM, Waldorf HA. A review of onabotulinumtoxinA (Botox). Aesthet Surg J. 2013 Mar;33(1 Suppl):9S-12S. doi: 10.1177/1090820X12474629. PMID 23515199
- [Background] Knopp MV, Balzer T, Esser M, Kashanian FK, Paul P, Niendorf HP. Assessment of utilization and pharmacovigilance based on spontaneous adverse event reporting of gadopentetate dimeglumine as a magnetic resonance contrast agent after 45 million administrations and 15 years of clinical use. Invest Radiol. 2006 Jun;41(6):491-9. doi: 10.1097/01.rli.0000209657.16115.42. PMID 16763467
- [Background] Montagna P. Migraine genetics. Expert Rev Neurother. 2008 Sep;8(9):1321-30. doi: 10.1586/14737175.8.9.1321. PMID 18759544
- [Background] Robbins MS, Lipton RB. The epidemiology of primary headache disorders. Semin Neurol. 2010 Apr;30(2):107-19. doi: 10.1055/s-0030-1249220. Epub 2010 Mar 29. PMID 20352581
- [Background] Levy D, Strassman AM, Burstein R. A critical view on the role of migraine triggers in the genesis of migraine pain. Headache. 2009 Jun;49(6):953-7. doi: 10.1111/j.1526-4610.2009.01444.x. PMID 19545256
- [Background] Cousins G, Hijazze S, Van de Laar FA, Fahey T. Diagnostic accuracy of the ID Migraine: a systematic review and meta-analysis. Headache. 2011 Jul-Aug;51(7):1140-8. doi: 10.1111/j.1526-4610.2011.01916.x. Epub 2011 Jun 7. PMID 21649653
- [Background] Olesen J, Burstein R, Ashina M, Tfelt-Hansen P. Origin of pain in migraine: evidence for peripheral sensitisation. Lancet Neurol. 2009 Jul;8(7):679-90. doi: 10.1016/S1474-4422(09)70090-0. PMID 19539239
- See also: Click here for more information about this study ASIS for Botox in Chronic Migraine — http://www.asis-inc.com